CLINICAL TRIAL: NCT00716092
Title: A 4-week, Randomized, Double Blind, Double Dummy, Placebo Controlled, Parallel Group Study Comparing the Influence of BI 1356 (5 mg) and Sitagliptin (100 mg) Administered Orally Once Daily on Various Biomarkers in Type 2 Diabetic Patients
Brief Title: The Effect of Linagliptin (BI 1356) on 24h-glucose Control and Various Biomarkers in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.37; 2007-007865-19 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Results first posted 2011-06-15 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; Sitagliptin Phosphate

ARMS (3):
- Placebo (Placebo Comparator): Patients received placebo matching 5mg linagliptin and placebo matching 100mg sitagliptin.
  Interventions: Drug: Placebo (linagliptin); Drug: Placebo (sitagliptin)
- Linagliptin (Experimental): Patients received 5mg linagliptin, and placebo matching 100mg sitagliptin.
  Interventions: Drug: Placebo (sitagliptin); Drug: Linagliptin
- Sitagliptin (Active Comparator): Patients received 100mg sitagliptin, and placebo matching 5mg linagliptin.
  Interventions: Drug: Placebo (linagliptin); Drug: Sitagliptin

INTERVENTIONS:
Drug: Placebo (linagliptin) — once daily for 28 days
  Arms: Sitagliptin
Drug: Placebo (linagliptin) — once daily for 28 days
  Arms: Placebo
Drug: Sitagliptin — 100 mg once daily for 28 days
  Arms: Sitagliptin
Drug: Placebo (sitagliptin) — once daily for 28 days
  Arms: Linagliptin
Drug: Placebo (sitagliptin) — once daily for 28 days
  Arms: Placebo
Drug: Linagliptin — 5mg once daily for 28 days
  Arms: Linagliptin

SUMMARY:
The objective of this study is to investigate the effect of BI 1356 on 24-h glucose control and various pharmacodynamic parameters in type 2 diabetic patients with inadequate glycaemic control.

ELIGIBILITY:
Inclusion criteria:

* Male and female patients with a diagnosis of type 2 diabetes mellitus and previously treated with not more than one drug
* Glycosylated haemoglobin A1 (HbA1c) 6.5 to 10.0% at Start of Run-in

Exclusion criteria:

* Myocardial infarction, stroke or transient ischemic attack "TIA" within 6 months prior to informed consent
* Impaired hepatic function
* Renal insufficiency with a creatinine clearance < 50 mL/min
* Treatment with rosiglitazone, pioglitazone, glucagon like peptide 1 (GLP-1) analogues, insulin, dipeptidyl peptidase 4 (DPP-4) inhibitors or anti-obesity drugs 3 months prior to informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2008-07; Primary Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- Germany (3):
  - 1218.37.49003 Boehringer Ingelheim Investigational Site, Berlin
  - 1218.37.49002 Boehringer Ingelheim Investigational Site, Mainz
  - 1218.37.49001 Boehringer Ingelheim Investigational Site, Neuss

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients randomized to receive treatment with matching placebo
- BI1356: Patients randomized to receive treatment with BI1356 5 mg
- Sitagliptin: Patients randomized to receive treatment with Sitagliptin 100 mg
Period: Overall Study
Arm/Group | Placebo | BI1356 | Sitagliptin
Started | 40 | 40 | 41
Completed | 38 | 39 | 41
Not Completed | 2 | 1 | 0
Not completed — Other incl. Lack of Efficacy | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI1356 | Sitagliptin | Total
Number analyzed (Participants) | 40 | 40 | 41 | 121
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (9.5) | 60.7 (10.11) | 62.0 (7.85) | 61.1 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 9 | 35
  Male | 29 | 25 | 32 | 86
Body Mass Index (BMI) continuous [Mean (Standard Deviation); unit: kg/m^2] | 30.3 (3.83) | 31.4 (4.48) | 30.7 (4.56) | 30.8 (4.29)
Glycosylated Hemoglobin A1 (HbA1C) continuous [Mean (Standard Deviation); unit: Percent] | 7.47 (0.53) | 7.32 (0.59) | 7.17 (0.44) | 7.32 (0.53)
Fasting plasma glucose (FPG) continuous [Mean (Standard Deviation); unit: mg/dL] | 172.8 (28.81) | 166.9 (27.65) | 160.3 (25.35) | 166.6 (27.55)

OUTCOME MEASURES:

1. Primary Outcome: Weighted Mean Glucose (WMG) Change From Baseline at Day 28
Description: The change from baseline reflects the day 28 WMG value minus the baseline WMG value. Means are treatment adjusted for baseline HbA1c, previous anti-diabetic medication, and baseline WMG.
Time Frame: Baseline and day 28
Population: The pharmacodynamic set(PD-set) consisted of all randomised patients who were treated with at least one dose of study drug. This analysis was based upon model with only BI 1356 and Placebo groups, further restricted to patients who had a baseline and at least one on-treatment value for WMG. Sitagliptin results are from model containing all 3 groups
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | BI1356 | Sitagliptin
Number analyzed (Participants) | 38 | 39 | 40
mg/dL | 0.1 (3.0) | -19.8 (2.9) | -26.1 (2.8)
Statistical Analysis 1: Comparison: Placebo vs BI1356; BI1356 minus Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — There was no adjustment for multiple primary endpoints, however a hierarchy approach to control for the Type-I error was used. If the endpoint WMG was not successful, any analysis of the GLP-1 (AUEC 0-24h) was to be considered descriptive; The primary analyses are based upon a model containing only BI1356 and Placebo. Sitagliptin values come from a different model containing all 3 groups; Mean Difference (Final Values) = -19.9, 95% CI [-28.0 to -11.9], Standard Error of Mean 4.0

2. Primary Outcome: GLP-1 (Glucagon Like Peptide 1) AUEC (0-2h) (Area Under Effect Curve) Change From Baseline at Day 28
Description: The change from baseline reflects the day 28 GLP-1 AUEC (0-2h) value minus the baseline GLP-1 AUEC (0-2h) value. Means are treatment adjusted for baseline HbA1c, previous anti-diabetic medication and baseline GLP-1.
Time Frame: Baseline and day 28
Population: The pharmacodynamic set(PD-set) consisted of all randomised patients who were treated with at least one dose of study drug. Analysis was based upon model with only BI 1356 and Placebo groups, further restricted to patients who had a baseline and at least one ontreatment value for GLP-1. Sitagliptin results are from model containing all 3 groups.
Measure: Mean (Standard Error); unit: pmol*h/L
Arm/Group | Placebo | BI1356 | Sitagliptin
Number analyzed (Participants) | 38 | 39 | 41
pmol*h/L | 0.4 (2.1) | 18.5 (2.1) | 15.3 (2.0)
Statistical Analysis 1: Comparison: Placebo vs BI1356; BI1356 minus Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — There was no adjustment for multiple primary endpoints, however a hierarchy approach to control for the Type-I error was used. If the endpoint WMG was not successful, any analysis of the GLP-1 (AUEC 0-24h) will be considered descriptive; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 18.1, 95% CI [12.4 to 23.9], Standard Error of Mean 2.9

3. Secondary Outcome: Fasting Plasma Glucose (FPG) Change From Baseline at Day 28
Description: The change from baseline reflects the day 28 FPG value minus the baseline FPG value. Means are treatment adjusted for baseline HbA1c, previous anti-diabetic medication and baseline FPG.
Time Frame: Baseline and day 28
Population: The pharmacodynamic set(PD-set) consisted of all randomised patients who were treated with at least one dose of study drug. This analysis was based upon model with only BI 1356 and Placebo groups, further restricted to patients who had a baseline and at least one on-treatment value for FPG. Sitagliptin results are from model containing all 3 groups
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | BI1356 | Sitagliptin
Number analyzed (Participants) | 38 | 39 | 41
mg/dL | -0.1 (3.6) | -10.9 (3.5) | -15.6 (3.1)
Statistical Analysis 1: Comparison: Placebo vs BI1356; BI1356 minus Placebo; Test type: Superiority or Other; p = 0.0283, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.8, 95% CI [-20.4 to -1.2], Standard Error of Mean 4.8

4. Secondary Outcome: Plasma Glucose Area Under Effect Curve (AUEC) (0-3h) Change From Baseline at Day 28
Description: The change from baseline reflects the day 28 Glucose AUEC (0-3h) value minus the baseline Glucose AUEC (0-3h) value. Means are treatment adjusted for baseline HbA1c, previous anti-diabetic medication and baseline plasma glucose AUEC (0-3h).
Time Frame: Baseline and day 28
Population: The pharmacodynamic set (PD-set) consisted of all randomised patients who were treated with at least one dose of study drug. This analysis was based upon model with only BI 1356 and Placebo, further restricted to patients who had a baseline and at least one on-treatment value for Glucose AUEC(0-3h). Sitagliptin results from model with all 3 groups.
Measure: Mean (Standard Error); unit: mg*h/dL
Arm/Group | Placebo | BI1356 | Sitagliptin
Number analyzed (Participants) | 38 | 39 | 41
mg*h/dL | 8.1 (15.1) | -98.4 (14.7) | -119.1 (13.3)
Statistical Analysis 1: Comparison: Placebo vs BI1356; BI1356 minus Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -106.5, 95% CI [-147.0 to -66.0], Standard Error of Mean 20.3

5. Other Pre Specified Outcome: Exploratory Sensitivity Analysis of the WMG Change From Baseline at Day 28
Description: The change from baseline reflects the day 28 WMG value minus the baseline WMG value. Means are treatment adjusted for baseline HbA1c, previous anti-diabetic medication and baseline WMG.
Time Frame: Baseline and day 28
Population: This analysis was based upon the PD-set further restricted to patients who had a baseline and at least one on-treatment value for WMG.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | BI1356 | Sitagliptin
Number analyzed (Participants) | 38 | 39 | 40
mg/dL | -0.2 (2.9) | -20.1 (2.8) | -26.1 (2.8)
Statistical Analysis 1: Comparison: BI1356 vs Sitagliptin; BI 1356 minus Sitagliptin. This analysis comparing BI1356 to Sitagliptin was conducted as an exploratory analysis at the time of analysing the study data. The study was not powered for such a comparison; Test type: Superiority or Other; p = 0.1274, ANCOVA; These measured values and statistical analysis come from a mixed model containing all three treatment groups, and adjusted as already described; Mean Difference (Final Values) = 6.0, 95% CI [-1.7 to 13.8], Standard Error of Mean 3.9

6. Other Pre Specified Outcome: Exploratory Sensitivity Analysis of GLP-1 AUEC (0-2h) Change From Baseline at Day 28
Description: as for outcome 2
Time Frame: Baseline and day 28
Population: This analysis was based upon the PD-set further restricted to patients who had a baseline and at least one on-treatment value for GLP-1.
Measure: Mean (Standard Error); unit: pmol*h/L
Arm/Group | Placebo | BI1356 | Sitagliptin
Number analyzed (Participants) | 38 | 39 | 41
pmol*h/L | -0.1 (2.0) | 18.1 (2.0) | 15.3 (2.0)
Statistical Analysis 1: Comparison: BI1356 vs Sitagliptin; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.3130, ANCOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 2.8, 95% CI [-2.7 to 8.2], Standard Error of Mean 2.7

7. Other Pre Specified Outcome: Exploratory Sensitivity Analysis of FPG Change From Baseline at Day 28
Description: as for outcome 3
Time Frame: Baseline and day 28
Population: This analysis was based upon the PD-set further restricted to patients who had a baseline and at least one on-treatment value for FPG.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | BI1356 | Sitagliptin
Number analyzed (Participants) | 38 | 39 | 41
mg/dL | 0.4 (3.2) | -10.3 (3.1) | -15.6 (3.1)
Statistical Analysis 1: Comparison: BI1356 vs Sitagliptin; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.2281, ANCOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 5.2, 95% CI [-3.3 to 13.8], Standard Error of Mean 4.3

8. Other Pre Specified Outcome: Exploratory Sensitivity Analysis of Plasma Glucose AUEC (0-3h) Change From Baseline at Day 28
Description: as for outcome 3
Time Frame: Baseline and day 28
Population: This analysis was based upon the PD-set further restricted to patients who had a baseline and at least one on-treatment value for Plasma Glucose AUEC (0-3h).
Measure: Mean (Standard Error); unit: mg*h/dL
Arm/Group | Placebo | BI1356 | Sitagliptin
Number analyzed (Participants) | 38 | 39 | 41
mg*h/dL | 9.8 (14.0) | -96.4 (13.5) | -119.1 (13.3)
Statistical Analysis 1: Comparison: BI1356 vs Sitagliptin; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.2230, ANCOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 22.7, 95% CI [-14.0 to 59.5], Standard Error of Mean 18.6

ADVERSE EVENTS:
Time Frame: From day of first dose until 7 days after last dose, up to 35 days
Arm/Group | Placebo | BI1356 | Sitagliptin
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 5/40 | 5/40 | 6/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=40) | BI1356 (N=40) | Sitagliptin (N=41)
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Headache (Nervous system disorders) | 3 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.